CLINICAL TRIAL: NCT04922255
Title: Pilot Trial of Non-Surgical Management for Women With Cystic Fibrosis and Urinary Incontinence
Brief Title: Cystic Fibrosis and Urinary Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We exhausted all ability to recruit from our study sites
Sponsor: Megan Bradley (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Megan Bradley, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21010012
Record Dates: First submitted 2021-05-17; First posted 2021-06-10 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence; Cystic Fibrosis
MeSH Terms: conditions — Urinary Incontinence; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- disposable urethral support device (Active Comparator): disposable urethral support device
  Interventions: Device: Disposable urethral support
- Reusable Underwear (Active Comparator): Reusable Underwear
  Interventions: Device: Reusable Underwear
- pelvic floor muscle therapy (PFMT) (Active Comparator): Pelvic floor muscle therapy
  Interventions: Behavioral: Pelvic floor physical therapy

INTERVENTIONS:
Device: Reusable Underwear — Reusable Underwear are similarly available for purchase online and are absorbent underwear for bladder leak protection
  Arms: Reusable Underwear
Device: Disposable urethral support — The disposable urethral support is a tampon-like device that is available over the counter to help women with urinary incontinence (UI)
  Arms: disposable urethral support device
Behavioral: Pelvic floor physical therapy — Experienced pelvic health physical therapists (at University of Pittsburgh) will complete two visits one week apart.
  Arms: pelvic floor muscle therapy (PFMT)

SUMMARY:
Evaluate the feasibility of a randomized controlled trial of non-surgical urinary incontinence (UI) management options for women with CF. The investigators will complete a pilot, feasibility study (n=30) to compare tolerability and symptom relief in women with CF and UI. Subjects will be recruited from the University of Pittsburgh Cystic Fibrosis Center after demonstrating bother from UI on initial phone script. Participants will undergo UI questionnaires and undergo a pelvic examination, non-invasive bladder scan ultrasound and a provocative stress test and then be randomized to either a disposable urethral support device (Impressa®), an absorbent product (Speax Reusable Underwear), or Pelvic floor muscle therapy. The primary outcome will be to determine the feasibility and tolerability of these options.

Hypothesis: All three non-surgical UI management options for women are feasible (as measured by 80% adherence to treatment assignment over 7 days) and tolerable (as measured by patient report via questionnaire).

The results from the proposed aims will provide important information about the experiences and symptom burden of women with CF and UI. Importantly, the investigators will also be able to answer the important questions of "Can it work?" and "Does it work?" as the investigators seek to construct the definitive, adequately powered trial of these therapies in women with CF and UI.

DETAILED DESCRIPTION:
Study Procedures: Participants will be recruited at routine cystic fibrosis (CF) clinic visits and via telephone screening. The investigators will again utilize the ISI for screening procedures with subjects required to have at incontinence at least as frequent as 'less than once a month' and at least as 'drops' to be eligible for enrollment. Informed consent will be obtained before any study procedures are initiated. Initial demographic questions and the King's Health Questionnaire (KHQ) will be completed at the baseline visit. Subjects will be given materials to complete a 2-day bladder diary. The bladder diary has participants track what they take in (fluids) and also their voided volumes throughout the day and night. Subjects will be given a hat to void in a collect the numbers/volume of voids and also leakage episodes. Pregnancy will be excluded by self-report. Participants will then have a pelvic exam for a visual urethral mobility examination and assessment of pelvic floor muscle strength to be completed by the principal investigator. The principal investigator will additionally first perform a bladder scan ultrasound to assess current bladder volume and then a cough stress test (CST). The exam will be performed in the supine/lithotomy position with ≥300 mL of fluid in the bladder. The investigators will have the subject cough forcefully 1-4 times and the examiner will directly visualize the urethral meatus for the presence of leakage. Leakage of fluid from the urethral meatus coincident with/simultaneous to the cough(s) is considered a positive test consistent with stress urinary incontinence (SUI).

Randomized feasibility trial (Table 2). At the baseline visit, women will be given a brief description of the three different treatment options and be initially asked to rank initial choice for treatment. Participants will then be randomized to either a disposable urethral support device (Impressa®), Speax™ Reusable Underwear, or pelvic floor muscle therapy (PFMT). Randomization will be in a 1:1:1 allocation without stratification by incontinence severity. The disposable Impressa® urethral support is a tampon-like device that is available over the counter to help women with urinary incontinence (UI). Speax Reusable Underwear are similarly available for purchase online and are absorbent underwear for bladder leak protection. Both the Impressa and Speax are commercially available and the Impressa is FDA approved. The Speax underwear are not a FDA regulated product. Urethral support device cohort - A week supply of the Impressa device will be provided and participants will be asked to complete a daily bladder diary for a total of 7 days. The instructions for use booklet will be provided. Subjects will be told that they can continuously utilize one Impressa for up to 12 hours. The investigators will ask subjects to wear for at least 12 hours a day but up to 24 if they desire. Reusable absorbent pad cohort - Three pairs of Speax underwear will be provided and subjects will complete a similar daily UI diary for 7 days. Subjects will be instructed to wear one pair of speax daily and may wash as they desire. Subjects will be provided the website for the product and The investigators will allow them to order whatever pair/size the subject desires. https://www.shethinx.com/pages/speax. PFMT cohort - Experienced pelvic health physical therapists (at both University of Pittsburgh) will complete two visits one week apart. Each PFMT visit will take ~60 minutes. The investigators will develop a standardized pelvic floor exercise intervention based on previous RCT for PFMT in women with MUI. The intervention will comprise: 1) Bladder training and delayed voiding techniques 2) Urgency suppression 3) SUI strategies (e.g., 'knack') and 4) Pelvic floor muscle (PFM) training for those agreeable to internal exams. The investigators will utilize Diaphragmatic breathing, Happy Baby Stretch with pelvic floor muscle (PFM) relaxation and lower abdominal myofascial release (MFR) to start. These are all non-internal stretching type exercises similar to yoga and will be performed for ~20-30 minutes. If the subject is willing the investigators will consider internal pelvic floor muscle training which will involve the physical therapist inserting one digit into the vagina in order to aid in muscle coordination. This will also be done for 20-30 minutes.

Subjects will not be blinded to their group assignment given the nature of the differences in management options. At the end of the treatment assignment all subjects will repeat the KHQ and a patient global impression of improvement (PGI-I). The PGI-I is a validated one question measure rating their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better) to 7 (Very much worse). All subjects will complete the follow-up questionnaires 7-days after the beginning of their assigned therapy.

Given the opportunity to gather acceptability on these options for a sensitive issue, subjects will be offered an option to further participate in one alternate therapy of their choosing. If subjects select this option, investigators will organize an additional week of therapy. Participants will only have to complete a BSW questionnaire and another PGI-I at the end of therapy. This is an option for all women in the study even if they initially had been randomized to their preferred option as participants may ultimately have not really liked that choice.

Acceptability and Feasibility assessment: Urethral support device cohort and Reusable absorbent pad cohort: Feasibility will be evaluated through assessment of use and product performance. Logs regarding utilization of assigned product will be completed daily. Patient treatment preference will be assessed after completion of both therapies utilizing the product performance questionnaire (PPQ). The PPQ is a 13-item product questionnaire that consists of product questions that are specific to incontinence products and includes questions about overall impression of product, ability to hold urine, ability to prevent odor, fit, discreteness, comfort when wet and dry, and ability to keep skin dry. PFMT cohort: Feasibility will be evaluated through assessment of adherence and self-reported success with ability to perform exercises. Adherence to intervention sessions will be documented by physical therapist using attendance logs. Adherence to home practice will be documented by participants in home logs that included the dates and times of practice. At the end of each physical therapy visit, participants will be asked to rate their confidence in performing the PFMT exercises featured in their program (extremely, very, moderately, somewhat, and not at all confident).

At the end of the study, all participants will be asked to indicate how easy it would be to continue practicing their assignment intervention (extremely, very, moderately, somewhat, and not at all easy). All subjects will complete a Benefit, Satisfaction, and Willingness to Continue (BSW) questionnaire. The investigators will consider therapy feasible (as measured by 80% adherence to treatment assignment over 7 days) and tolerable (as measured by patient report via questionnaire). By allowing subjects to choose another one of the arms after their randomization this will give us further, important information about feasibility and patient preference for a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 years or older
* Diagnosis of CF
* Self-reported UI (at least answer of "a little" on King's Health Questionnaire - Question #2)
* Fluent in spoken English
* Ability to present for in-office exam and study procedures

Exclusion Criteria:

* Age <18 years
* No UI
* Inability to comply with study protocol
* No diagnosis of Cystic Fibrosis
* Pregnant

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 15 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Bradley, MD, Principal Investigator — University of Pittsbugh School of Medicine
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Started | 4 | 6 | 5
Completed | 4 | 4 | 4
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT) | Total
Number analyzed (Participants) | 4 | 6 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.7) | 42.6 (17.9) | 34.8 (16.7) | 37.3 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 15
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 4 | 6 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Improvement-Incontinence
Description: The Patient Global Impression of Improvement-Incontinence (PGI-I) is a validated one question measure rating their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better) to 7 (Very much worse). It is a score calculated at Day 7.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Number analyzed (Participants) | 4 | 4 | 4
score on a scale | 2.25 (0.05) | 3.00 (0.05) | 3.75 (0.05)
Statistical Analysis 1: Comparison: Disposable Urethral Support Device vs Reusable Underwear vs Pelvic Floor Muscle Therapy (PFMT); Test type: Superiority; p = 0.04, ANOVA

2. Secondary Outcome: Patient Treatment Preference
Description: Patient treatment preference will be assessed after completion of initial assigned therapy utilizing the product performance questionnaire (PPQ). The PPQ is a 13-item product questionnaire that consists of product questions that are specific to incontinence products and includes questions about overall impression of product, ability to hold urine, ability to prevent odor, fit, discreteness, comfort when wet and dry, and ability to keep skin dry. Patients are allowed to answer each question with either "unacceptable (1)," "acceptable (2) ," or "good (3) " to each question. Therefor minimum on questionnaire is a 0 and maximum is 39 with higher score showing improved patient treatment preference/performance of product.
Time Frame: 7 days
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Number analyzed (Participants) | 4 | 4 | 4
units on a scale | 23 [19 to 34] | 37 [31 to 38] | 38 [37 to 39]
Statistical Analysis 1: Comparison: Disposable Urethral Support Device vs Reusable Underwear vs Pelvic Floor Muscle Therapy (PFMT); Test type: Superiority; p = 0.50, Kruskal-Wallis

3. Secondary Outcome: King's Health Questionnaire
Description: The KHQ is a 21-item scale with 9 domains: general health perceptions, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, Sleep/Energy, and severity measures and an 11-item symptom severity score. (Hebbar et al., 2015)
  Each question has four options "not at all", "a little", "moderately" and "a lot". (numerically 1-4) The general health perception domain has five choices ("very good", "good", "fair", "bad" and "very bad") (numerically 1-5). The scores are then converted to "out of 100" with accepted formulas. For example for Q1 the overall score = ((actual score-1)/4)*100 In the KHQ, a minimum possible score of zero is assigned to the best health and a maximum possible score of 100 is assigned to the worst health. The 0-100 scale is used for each item and each subscale separately.
  You can then report a total average score across all domains which is reported here
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Number analyzed (Participants) | 4 | 4 | 4
units on a scale | 66.7 (23.6) | 33.3 (23.6) | 25 (14.4)
Statistical Analysis 1: Comparison: Disposable Urethral Support Device vs Reusable Underwear vs Pelvic Floor Muscle Therapy (PFMT); Test type: Superiority; p = 0.30, ANOVA

4. Secondary Outcome: Adherence Logs
Description: Subjects will be asked to document their adherence to therapy on a daily basis and outcome will be reported as the percentage of participants with 100% adherence (responded yes to adherence to therapy all 7 days of therapy on their daily log)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Number analyzed (Participants) | 4 | 4 | 4
Participants | 3 | 3 | 4
Statistical Analysis 1: Comparison: Disposable Urethral Support Device vs Reusable Underwear vs Pelvic Floor Muscle Therapy (PFMT); Test type: Superiority; p = 0.70, Chi-squared

5. Secondary Outcome: Benefits, Satisfaction, and Willingness to Continue
Description: At the end of the study, all participants will be asked to indicate how easy it would be to continue practicing their assignment intervention (extremely, very, moderately, somewhat, and not at all easy) and complete the Benefit, Satisfaction, and Willingness to Continue (BSW) questionnaire which asks "would you be willing to continue treatment with this product or therapy?" The reported outcome is the number of participants per group that answered "Yes" to this question.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
Number analyzed (Participants) | 4 | 4 | 4
Participants | 0 | 4 | 4
Statistical Analysis 1: Comparison: Disposable Urethral Support Device vs Reusable Underwear vs Pelvic Floor Muscle Therapy (PFMT); Test type: Superiority; p = 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 week
Description: Self-reported adverse events
Arm/Group | Disposable Urethral Support Device | Reusable Underwear | Pelvic Floor Muscle Therapy (PFMT)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT04922255/Prot_SAP_002.pdf